## Balance Recovery Training for Fall Prevention in Retirement Communities

NCT02551666

October 13, 2015

## STATISTICAL ANALYSIS PLAN

Baseline-post intervention changes in clinical and reactive balance measures were compared between RBT and Tai Chi groups using a mixed model (SAS PROC MIXED procedure, SAS Institute Inc., Cary NC) that accounted for fixed and random effects, and within-participant correlation. For the clinical tests, fixed effects of intervention (RBT or Tai Chi), time (one week, one month, three months, or six months post-intervention), and intervention\*time were included, as well as covariates of baseline (pre-intervention) performance, age, gender, and baseline reactive balance rating score. For the reactive balance measures, fixed effects of intervention, time, speed, and all two-factor interactions were included, along with the same covariates noted above. Hierarchical models were used in analyzing reactive balance measures to account for the two levels of repeated measures (time and speed) and the two replications of each time-speed combination. *A priori* simple effects investigated differences between intervention groups at each time point to address our hypotheses, and the Tukey-Kramer method was used to adjust for Type I error rate, with a significance level of  $p \le .05$ . Differences in categorical variables between groups were evaluated using Fisher's Exact Test.